CLINICAL TRIAL: NCT00163982
Title: Vasoactive Peptides in Portal Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AH4204
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2005-09

CONDITIONS: Portal Hypertension
Keywords: HVPG > 12 mmHg
MeSH Terms: conditions — Hypertension, Portal | interventions — Norfloxacin

INTERVENTIONS:
Drug: Norfloxacin

SUMMARY:
This study is looking at the detection of vasoactive peptides in portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* HVPG >= 12 mmHg

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William W Kemp, MBBS, FRACP, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia